CLINICAL TRIAL: NCT04395950
Title: A Phase 1B, Single-Blinded, Linear Two Period, Placebo-controlled Study to Evaluate the Effects of 10 mg/Day of PF-05221304, Liver Targeted Acetyl-CoA Carboxylase Inhibitor (ACCi) on Very Low Density Lipoprotein ApoB100 and TG Secretion
Brief Title: Effects of ACC Inhibitor on Lipid and Lipoprotein Metabolism
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAS9106
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: NASH (Nonalcoholic Steatohepatitis); NAFLD (Nonalcoholic Fatty Liver Disease)
Keywords: NASH; NAFLD; non-alcoholic steatohepatitis; liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-0522130 (Active Comparator): PF-05221304 10 mg daily (two 5mg tablets daily in the morning).
  Interventions: Drug: PF-05221304
- Placebo (Placebo Comparator): Placebo (two tablets daily in the morning).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05221304 — PF-05221304 10 mg daily (two 5mg tablets daily in the morning for 6 weeks)
  Other Names: PF1304
  Arms: PF-0522130
Drug: Placebo — Placebo two tablets daily in the morning for 6 weeks
  Other Names: Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of an investigational drug, PF-05221304 (PF'1304) on the way the liver handles fat. The planned study will identify why the fat in the blood increases at the same time this drug reduces fat in the liver. The study will have two treatment periods of 6 weeks each, separated by a 3 week rest period with no treatment. The subjects will receive the active drug in one of the 6 week treatment periods and a placebo in the other 6 week period. The investigators will know when the subjects are receiving active treatment or placebo, but the subject will not know.

DETAILED DESCRIPTION:
Nonalcoholic Fatty Liver Disease (NAFLD) is a condition in which fat builds up in the liver. As its name suggests, it is not associated to heavy alcohol use. Non-Alcoholic Steatohepatitis (NASH) is a condition of liver inflammation and damage that is caused by the buildup of fat in the liver. It is usually associated with prediabetes, diabetes (high blood sugar in the blood), a high concentration of fat (triglycerides) in the blood, and obesity (increase in fat all over the body). The signs and symptoms of NASH are often not seen until the liver is damaged beyond repair, making NASH very difficult to diagnose (be picked up by your doctor) in its early stages where treatments might be able to reverse the damage.

There are no treatments currently approved for people with NASH but several new medications are under study in people with NAFLD or NASH. This study uses a treatment being developed for treating NASH. The investigators will conduct a study to assess the effects of PF-05221304 (PF'1304) on the way the liver handles fat. In early studies, this new drug has shown promise for lowering the level of fat in the liver. However, it also, unexpectedly, increases the level of fat in the blood, which could increase the risk of heart disease and inflammation of the pancreas.

The planned study will identify why the fat in the blood increases. Subjects will undergo a screening period where we will obtain medical history and physical exam. Additionally, we will obtain the results of liver imaging or liver biopsy previously performed by the subject's doctor that confirm the presence of an abnormal amount of liver fat and liver stiffness. The enrolled subjects will receive placebo (an inactive pill) during the first 6 weeks, followed by a 3 week washout period and then 6 weeks of active treatment. Blood samples will be collected during outpatient visits to check for study safety and measurements of fat in the blood and particles that carry that fat. There will also be 2 long outpatient studies that last approximately 15 hours each, where we will test why there is increase in fat blood levels during treatment with PF'1304. All visits will occur at the CUIMC Irving Institute for Clinical and Translational Research. Subject risk will be minimized through strict eligibility criteria to avoid enrollment of unstable or high-risk subjects and by close monitoring of adverse events (AE's), laboratory parameters, and vital signs during the study. In addition, blood fat levels will be measured on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of ≥ 25 kg/m2 but < 40 kg/m2 and at least 2 of 5 traits of metabolic syndrome (fasting blood glucose >100 mg/dl or diagnosis of diabetes mellitus; BP >130/85; fasting TG >150 mg/dl; HDL cholesterol <40 mg/dl for men and <50 mg/dl for women; waist circumference >101 cm for men and >89 cm for women).
* NASH will be defined as a FibroScan® of CAP >280 db/m and >7 kPa, OR demonstrated by liver biopsy, plus:
* ALT > ULN but < 5 X ULN.
* FIB4 score <3.5 (see below)
* BP of ≤ 160/100 mmHg.
* Alkaline phosphatase ≤ ULN.
* Total bilirubin ≤ ULN (unless the subject has Gilbert's syndrome, a benign genetic problem where bilirubin is not conjugated normally and indirect bilirubin (unconjugated bilirubin increases) in which case direct bilirubin must be ≤ ULN with total bilirubin > ULN).
* Platelet count ≥ LLN (155,000/mm3).
* Albumin ≥ LLN (3.0 g/L).
* INR ≤ 1.3.
* Fasting serum triglycerides ≤ 350 mg/dL either non-pharmacologically managed or pharmacologically managed with stable doses of up to 3 oral agents for at least 6 months. They may be receiving statins if the dose has been stable for at least 3 months.
* Subjects may have diabetes but must have an HbA1C ≤ 8.0% with glycemic control either non-pharmacologically managed or pharmacologically managed with stable doses of up to 3 oral agents for at least 6 months. Subjects taking a stable dose of long-acting insulin or an injectable GLP-1 inhibitor may be enrolled at the discretion of the investigators.
* No changes in drugs affecting blood lipid or glucose or insulin levels will be permitted during the study without approval by the investigators.

Exclusion Criteria:

* Individuals with a history of plasma TG >1000 mg/dl and/or pancreatitis.
* Females of childbearing potential.
* Chronic kidney disease defined by estimated glomerular filtration rate < 30 ml/min/1.73 m² by the modification of diet in renal disease equation.
* Documented chronic hepatitis B or C. Subjects with hepatitis C are eligible provided there is proof of sustained virology response (SVR) for ≥ 3 years.
* History of active malignancy within 5 years (subjects with non-melanoma skin cancer may be included).
* Any other disease, condition, or laboratory value that, in the opinion of the principal investigator or clinical study team would place the subject at an unacceptable risk or interfere with the evaluation of the investigative product.
* History of organ transplantation (other than corneal).
* History of hepatobiliary malignancy even if subject "cured".
* Pancreas divisum or a congenital abnormality of the pancreas
* History of pancreatic surgery.
* Subjects taking anti -coagulants or anti-platelet agents other than 81 mg ASA daily.
* Treatment with immunomodulators.
* Drugs associated with acute pancreatitis as asparaginase, azathioprine, didanosine, mecaptourinol, mesalamine, opiates, pentamidine, pentavalent anti-monials, valproic acid, and rifampin.
* OATP inhibitors such as gemfibrozil and cyclosporinea. Drugs substrates for CYP3A4/5 with a narrow therapeutic index - these include: alfentanil, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, and terfenadine will be reason for exclusion.

a = the major clearance mechanism of PF-05221304 is active uptake into liver (mainly via hepatic transporters OATP1B1/1B3) followed by hepatic carbonyl reductase 1, 11b-hydroxysteroid dehydrogenase, and CYP 3A4/5-mediated metabolism. It is anticipated that potent OATP inhibitors may increase plasma concentrations of PF-05221304. As such, subjects treated with clinically relevant OATP inhibitors will be excluded from this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Rate of Secretion (also called production-PR) of VLDL TG (mg/kg/day) | Up to 20 weeks
  This is also called the production rate of very low density lipoprotein (VLDL) triglycerides (TG).
Fractional Clearance Rate (FCR) of VLDL TG (pool/day) | Up to 20 weeks
  This is obtained from the modeling of enrichment data obtained by mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ginsberg, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi SH, Ginsberg HN. Increased very low density lipoprotein (VLDL) secretion, hepatic steatosis, and insulin resistance. Trends Endocrinol Metab. 2011 Sep;22(9):353-63. doi: 10.1016/j.tem.2011.04.007. Epub 2011 May 26. PMID 21616678
- [Background] Donnelly KL, Smith CI, Schwarzenberg SJ, Jessurun J, Boldt MD, Parks EJ. Sources of fatty acids stored in liver and secreted via lipoproteins in patients with nonalcoholic fatty liver disease. J Clin Invest. 2005 May;115(5):1343-51. doi: 10.1172/JCI23621. PMID 15864352
- [Background] Diraison F, Moulin P, Beylot M. Contribution of hepatic de novo lipogenesis and reesterification of plasma non esterified fatty acids to plasma triglyceride synthesis during non-alcoholic fatty liver disease. Diabetes Metab. 2003 Nov;29(5):478-85. doi: 10.1016/s1262-3636(07)70061-7. PMID 14631324
- [Background] Kim CW, Addy C, Kusunoki J, Anderson NN, Deja S, Fu X, Burgess SC, Li C, Ruddy M, Chakravarthy M, Previs S, Milstein S, Fitzgerald K, Kelley DE, Horton JD. Acetyl CoA Carboxylase Inhibition Reduces Hepatic Steatosis but Elevates Plasma Triglycerides in Mice and Humans: A Bedside to Bench Investigation. Cell Metab. 2017 Aug 1;26(2):394-406.e6. doi: 10.1016/j.cmet.2017.07.009. PMID 28768177
- [Background] Goedeke L, Bates J, Vatner DF, Perry RJ, Wang T, Ramirez R, Li L, Ellis MW, Zhang D, Wong KE, Beysen C, Cline GW, Ray AS, Shulman GI. Acetyl-CoA Carboxylase Inhibition Reverses NAFLD and Hepatic Insulin Resistance but Promotes Hypertriglyceridemia in Rodents. Hepatology. 2018 Dec;68(6):2197-2211. doi: 10.1002/hep.30097. PMID 29790582
- [Background] Reyes-Soffer G, Moon B, Hernandez-Ono A, Dionizovik-Dimanovski M, Jimenez J, Obunike J, Thomas T, Ngai C, Fontanez N, Donovan DS, Karmally W, Holleran S, Ramakrishnan R, Mittleman RS, Ginsberg HN. Complex effects of inhibiting hepatic apolipoprotein B100 synthesis in humans. Sci Transl Med. 2016 Jan 27;8(323):323ra12. doi: 10.1126/scitranslmed.aad2195. PMID 26819195
- [Background] Ramakrishnan R, Ramakrishnan JD. Using mass measurements in tracer studies--a systematic approach to efficient modeling. Metabolism. 2008 Aug;57(8):1078-87. doi: 10.1016/j.metabol.2008.03.011. PMID 18640385
- [Background] Hellerstein MK, Neese RA. Mass isotopomer distribution analysis at eight years: theoretical, analytic, and experimental considerations. Am J Physiol. 1999 Jun;276(6):E1146-70. doi: 10.1152/ajpendo.1999.276.6.E1146. PMID 10362629
- [Background] Caulfield MP, Li S, Lee G, Blanche PJ, Salameh WA, Benner WH, Reitz RE, Krauss RM. Direct determination of lipoprotein particle sizes and concentrations by ion mobility analysis. Clin Chem. 2008 Aug;54(8):1307-16. doi: 10.1373/clinchem.2007.100586. Epub 2008 May 29. PMID 18515257